CLINICAL TRIAL: NCT02372123
Title: The Effect of Connective Tissue Massage in Women With Primary Dysmenorrhoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SERAP KAYA, project manager, Hacettepe University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GO15/98
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Dysmenorrhea; Pelvic Pain
Keywords: Dysmenorrhea; Primary dysmenorrhea; physiotherapy; massage; connective tissue massage; connective tissue manipulation
MeSH Terms: conditions — Dysmenorrhea; Pelvic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Other): lifestyle advice
  Interventions: Other: lifestyle advice
- intervention (Active Comparator): connective tissue manipulation
  Interventions: Other: lifestyle advice; Other: connective tissue manipulation

INTERVENTIONS:
Other: lifestyle advice — Investigators will give lifestyle advice to patients such as exercising regularly, limiting caffeine, sugar and alcohol intake, reduction or cessation of smoking
Other: connective tissue manipulation — Investigators will apply connective tissue manipulation on lumbosacral, lower thoracic, and anterior pelvic regions starting from the estimated time of ovulation until the next period begins
  Arms: intervention

SUMMARY:
The aim of this study is to investigate the effect of connective tissue manipulation on pain threshold in women with primary dysmenorrhoea. According to literature, there are studies that measure the pain threshold. But there is no randomized controlled trial which explore the short and long-term effects of connective tissue manipulation on primary dysmenorrhoea. Hypothesis of this study is that connective tissue manipulation increases pain threshold and decreases severity of pain in women suffer with primary dysmenorrhoea.

DETAILED DESCRIPTION:
Dysmenorrhoea has been defined painful menstruation. It is divided primary and secondary dysmenorrhoea according to the pathophysiology. Primary dysmenorrhoea is severe menstrual pain, occurs a short time after menarche and without pelvic pathology. Secondary dysmenorrhoea is severe menstrual pain that occurs related to pelvic pathology. In primary dysmenorrhoea, pain usually begins with menstruation and ends in 48-72 hours. Pain is usually felt in the lower abdomen and lumbosacral region. Fatigue, headache, vomiting, diarrhea and constipation may be accompanied by primary dysmenorrhoea.

It is difficult to determine the incidence and etiology of dysmenorrhoea because of the variety of the criteria used in the diagnosis of the dysmenorrhoea and subjective symptoms. But current studies show that primary dysmenorrhoea is common gynecological problem that affects majority of women. Tu et al. indicated that prevalence of primary dysmenorrhoea was between 20-90% percent and 15% of cases had severe symptoms.

Although the etiology of primary dysmenorrhoea is not fully understood, excessive prostaglandin production is believed to cause abnormal uterine activity. Hyperalgesia is present especially in the deep tissue during the menstrual cycle.

Various approaches have been proposed until now for the treatment of patients with dysmenorrhoea. These are medical treatments (for example paracetamol, NSAID, oral contraceptives), alternative treatments (for example herbal products and nutritional supplements, dietary changes), surgical treatments and physiotherapy and rehabilitation approaches. Connective tissue manipulation (CTM), physiotherapy and rehabilitation approach, has been found by German physiotherapist Elizabeth Dicke in 1929. CTM is a manual reflex therapy, which produces autonomic responses via cutaneous-visceral reflexes. This safe and effective technique consists short and long tractions, which performed on the patients' skin by the skilled and experienced physiotherapist. Although the effect mechanism of CTM has not been fully understood yet, it is known that the treatment method stimulates autonomic nervous system to rebalance the parasympathetic and sympathetic functions. CTM produces autonomic stimulus when the stroke is performed on the skin and blood vessels are stimulated by autonomic nerve endings located in the tissue interfaces. It has also found that stimulation of autonomic nerve endings may results in reduction of sympathetic vasoconstrictor tone leads to vasodilatation. Stimulation of skin with strokes affects segmental reflexes. It is known that stimulation of segmental reflexes can be used in treatment of organ dysfunctions. CTM applied to affected dermatome generates reflex effects in the associated organs, provides healing by increasing circulation and decreasing pain. Skin alterations and subcutaneous tissue tension are observed in the dermatomes and myotomes, which are innervated by same spinal cord level with malfunctioning organ. In addition to these effects, powerful stimulation of cutaneous mechanoreceptor induces gate control mechanism, increases pain threshold and decreases stress hormones and muscle tension.

The aim of this study is to investigate the effect of connective tissue manipulation on pain threshold in women with primary dysmenorrhoea. According to literature, there are studies that measure the pain threshold. But there is no randomized controlled trial which explore the short and long-term effects of connective tissue manipulation on primary dysmenorrhoea. Hypothesis of this study is that connective tissue manipulation increases pain threshold and decreases severity of pain in women suffer with primary dysmenorrhoea.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women: aged over 18 years, diagnosis of primary dysmenorrhea according to Primary Dysmenorrhea Consensus Guideline, having regular menstrual cycles, a history of menstrual pain starting in the first few years after menarche and menstrual pain rated higher than 40 mm on a visual analog scale considering the last six months

Exclusion Criteria:

* Menstrual pain below 40 mm on the VAS
* Severe gastrointestinal, urogynecological or autoimmune disease
* other chronic pain syndromes
* psychiatric disorder
* childbirth
* positive pregnancy test
* intrauterine device
* urogynecologic surgery
* chronic medication including oral contraceptives or antidepressants for at least six months prior to study
* irregular menstrual cycles
* a history or ultrasonographic observation of pathologic conditions

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
menstrual pain intensity | one month

SECONDARY OUTCOMES:
Menstrual Attitude Score | one month
Number of pain medication | one month
Menstrual Symptom Score | one month
Menstrual Pain Catastrophizing Score | one month

OTHER OUTCOMES:
treatment satisfaction score | one month
compliance with advices | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Arendt-Nielsen L, Madsen H, Jarrell J, Gregersen H, Drewes AM. Pain evoked by distension of the uterine cervix in women with dysmenorrhea: evidence for central sensitization. Acta Obstet Gynecol Scand. 2014 Aug;93(8):741-8. doi: 10.1111/aogs.12403. Epub 2014 May 24. PMID 24773180
- [Result] Molins-Cubero S, Rodriguez-Blanco C, Oliva-Pascual-Vaca A, Heredia-Rizo AM, Bosca-Gandia JJ, Ricard F. Changes in pain perception after pelvis manipulation in women with primary dysmenorrhea: a randomized controlled trial. Pain Med. 2014 Sep;15(9):1455-63. doi: 10.1111/pme.12404. Epub 2014 Mar 25. PMID 24666560
- [Result] Tu CH, Niddam DM, Chao HT, Chen LF, Chen YS, Wu YT, Yeh TC, Lirng JF, Hsieh JC. Brain morphological changes associated with cyclic menstrual pain. Pain. 2010 Sep;150(3):462-468. doi: 10.1016/j.pain.2010.05.026. PMID 20705214
- [Result] Holey LA, Dixon J, Selfe J. An exploratory thermographic investigation of the effects of connective tissue massage on autonomic function. J Manipulative Physiol Ther. 2011 Sep;34(7):457-62. doi: 10.1016/j.jmpt.2011.05.012. Epub 2011 Jul 23. PMID 21875520
- [Result] Holey LA, Dixon J. Connective tissue manipulation: a review of theory and clinical evidence. J Bodyw Mov Ther. 2014 Jan;18(1):112-8. doi: 10.1016/j.jbmt.2013.08.003. Epub 2013 Sep 8. PMID 24411158
- [Result] Reed BV, Held JM. Effects of sequential connective tissue massage on autonomic nervous system of middle-aged and elderly adults. Phys Ther. 1988 Aug;68(8):1231-4. PMID 3399521
- [Result] As-Sanie S, Harris RE, Harte SE, Tu FF, Neshewat G, Clauw DJ. Increased pressure pain sensitivity in women with chronic pelvic pain. Obstet Gynecol. 2013 Nov;122(5):1047-1055. doi: 10.1097/AOG.0b013e3182a7e1f5. PMID 24104772
- [Result] Granot M, Yarnitsky D, Itskovitz-Eldor J, Granovsky Y, Peer E, Zimmer EZ. Pain perception in women with dysmenorrhea. Obstet Gynecol. 2001 Sep;98(3):407-11. doi: 10.1016/s0029-7844(01)01465-x. PMID 11530120